CLINICAL TRIAL: NCT05627414
Title: Clinical Study on the Efficacy and Safety of Disitamab Vedotin Combined With Sintilimab and S-1 in the Conversion Treatment of HER2 Overexpression Unresectable Gastric Cancer
Brief Title: Conversion Therapy of Disitamab Vedotin Combined With Sintilimab and S-1 in HER2 Overexpression Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20221046
Record Dates: First submitted 2022-11-17; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Gastric Cancer
Keywords: Conversion therapy; Disitamab Vedotin; HER2 overexpression
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; sintilimab; S 1 (combination); potassium oxonate; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin Combined With Sintilimab and S-1 (Experimental): 30 HER2 overexpression unresectable gastric cancer patients will enrolle and treate with Disitamab Vedotin, Sintilimab and S-1. During the study period, imaging examinations were conducted every 6-12 weeks to evaluate the tumor and whether it reached the operable standard. The scheme and duration of postoperative adjuvant treatment were determined by the investigator according to the patient's conditions (Sintilimab was recommended to be maintained for 1 year, and other drugs were increased or decreased according to the patient's conditions).
  Interventions: Drug: Disitamab Vedotin; Drug: Sintilimab; Drug: S-1; Procedure: Intraperitoneal chemotherapy with paclitaxel

INTERVENTIONS:
Drug: Disitamab Vedotin — 2.5mg/kg，IV，Q3W
  Other Names: RC48
Drug: Sintilimab — 200 mg，IV，Q3W
  Other Names: TYVYT
Drug: S-1 — 40~60mg / m2, bid, d1-14, repeated every 3 weeks.
  Other Names: Tegafur，Gimeracil and Oteracil Potassium Capsules
Procedure: Intraperitoneal chemotherapy with paclitaxel — Paclitaxel (PTX) was used with a dose of 60mg / m2, Q3W. （Only for patients with peritoneal metastases）
  Other Names: Paclitaxel (PTX)

SUMMARY:
This is a phase II, one-arm study, which is aiming to evaluate the feasibility of combination of Disitamab Vedotin, Sintilimab and S-1 as conversion therapy in patients with HER2 overexpression unresectable gastric cancer .

DETAILED DESCRIPTION:
In this study, 30 HER2 overexpression unresectable gastric cancer patients will enrolle and treate with Disitamab Vedotin, Sintilimab and S-1. During the study period, imaging examinations were conducted every 6-12 weeks to evaluate the tumor and whether it reached the operable standard. The scheme and duration of postoperative adjuvant treatment were determined by the investigator according to the patient's conditions (Sintilimab was recommended to be maintained for 1 year, and other drugs were increased or decreased according to the patient's conditions). During the study, safety evaluation and effectiveness evaluation will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 1) Volunteer to take part in the study ;
* 2) Age 18~70 (including 70), male or female;
* 3) Gastric cancer or adenocarcinoma of gastroesophageal junction confirmed by histology and/or cytology;
* 4) Has a single initial unresectable factor. For example, peritoneal metastasis (P1),Intraperitoneal free cancer cells positive (CY1), Paraaortic lymph node metastasis, liver metastasis (≤ 3 lesions, and ≤ 5 cm for a single lesion), ovarian metastasis;
* 5) Have not received systematic treatment;
* 6) The HER2 immunohistochemistry (IHC) test result is IHC 3+or 2+, and the previous test results of the subject (confirmed by the investigator) are acceptable;
* 7) At least one assessable lesion (RECIST 1.1 );
* 8) Expected survival time ≥ 6 months;
* 9) ECOG 0-1;
* 10) Major organs are functioning normally；

Exclusion Criteria:

* 1) Have a history of malignant tumors other than gastric cancer, except for the following two cases:

  1. The patient has received possible curative treatment and there is no evidence of the disease within 5 years;
  2. The resected skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ and other carcinoma in situ were successfully received;
* 2) Suffering from diseases that affect the absorption, distribution, metabolism or clearance of the study drug (such as severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorder, etc.);
* 3) Have received allogeneic stem cells or solid organ transplantation in the past;
* 4) Patients who have received other anti-tumor systemic therapy in the past (including traditional Chinese medicine with anti-tumor indications), and have been less than 4 weeks from the completion of treatment to the administration of this study, or the adverse events caused by previous treatment have not recovered to ≤ CTCAE level 1 (except hair loss and pigmentation);
* 5) Previous or current congenital or acquired immunodeficiency disease;
* 6) Active or previously recorded autoimmune diseases or inflammatory diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, hypophysitis, hyperthyroidism or hypothyroidism, asthma requiring bronchodilators, etc.), vitiligo or asthma that has completely alleviated in childhood, Those who do not need any intervention after adulthood can be included;
* 7) Systemic immunosuppressive drugs were used within 2 weeks before enrollment, or were expected to be required during the study, except for the following:

  d) Corticosteroids for intranasal, inhalation, external or local injection (such as intra-articular injection);

  e) The dose of prednisone or other equivalent systemic corticosteroids does not exceed 10 mg/day;

  f) Preventive use of corticosteroids for hypersensitivity;
* 8) Allergic to the study drug;
* 9) Thrombosis or thromboembolism events occurred in the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc;
* 10) Patients at risk for severe bleeding；
* 11) Cardiovascular diseases with significant clinical significance;
* 12) Other significant clinical and laboratory abnormalities, which the researchers think affect the safety evaluation;
* 13) Serious infection in active period or poorly controlled clinically;
* 14) Not recovered from the operation;
* 15) Pregnant or lactating women, and women or men with fertility who are unwilling or unable to take effective contraceptive measures;
* 16) Other situations that the investigator thinks are not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 1 year
  The proportion of patients who underwent R0 surgery among all patients.

SECONDARY OUTCOMES:
objective response rate (ORR) | up to one year
  The proportion of patients who achieved patial response and complete reponse per RECIST version 1.1.
overall survival (OS) | From the first dose to death from any cause, up to two years.
  median OS or OS rate
Recurrence free survival（RFS） | From the first dose to recurrence or death from any cause, up to two years.
  median RFS or RFS rate
safety profile | up to 30 days after last treatment administration
  The grade and proportion of adverse events, treatment related adverse events, immune-related adverse events (irAEs), serious adverse events, and perioperative complications, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, Master, Principal Investigator — ianjin Medical University Cancer Institute and Hospital